CLINICAL TRIAL: NCT04774614
Title: Shade Match, Marginal Adaptation and Patient Satisfaction of VITA ENAMIC multiColor Versus IPS e.Max CAD Anterior Laminate Veneers (Randomized Clinical Trial)
Brief Title: Shade Match, Marginal Adaptation and Patient Satisfaction of VITA ENAMIC multiColor Versus IPS e.Max CAD Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nancy Sayed Abdel Aziz Abdel Aal Khalil, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22 10 20
Record Dates: First submitted 2021-01-17; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Shade Match

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VITA ENAMIC multiColor anterior laminate veneers (Experimental)
  Interventions: Procedure: anterior laminate veneers
- IPS e.max CAD anterior laminate veneers (Active Comparator)
  Interventions: Procedure: anterior laminate veneers

INTERVENTIONS:
Procedure: anterior laminate veneers — VITA ENAMIC multiColor

SUMMARY:
It is assumed that there will be no difference in shade match, marginal adaptation and patient satisfaction between VITA ENAMIC multiColor and IPS e.max CAD anterior laminate veneers.

DETAILED DESCRIPTION:
Study settings:

This study will be carried out on patients enrolled from the Outpatient clinic in fixed prosthodontics clinic, Faculty of Oral and Dental Medicine, Cairo University.

Participant timeline:

The patient will be treated in visits designated as follows:

1. st Visit: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination and primary impression for diagnostic cast construction.
2. nd Visit: Teeth preparation, secondary impression and temporary restoration.
3. rd Visit : Try in
4. th Visit: Placement and permanent cementation of the final restoration. Shade match, marginal adaptation and patient satisfaction will be evaluated immediately after cementation

Data collection methods

Primary outcome (Shade match) will be assessed by using Modified United State Public Health Service Criteria (Modified USPHS Criteria).

Secondary outcomes:

Marginal adaptation will be assessed by modified USPHS criteria. Patient's satisfaction will be assessed using nominal scores (non-acceptable, acceptable, good and excellent).

Data management:

All data will be entered electronically in an Excel sheet. Patient files are to be stored in numerical order in a secured place.

Statistical methods:

* All Data will be collected, checked, revised, tabulated and entered into the computer.
* Data will be analyzed using IBM advance statistics (Statistics package for social sciences) version 21 (SPSS inc, Chicago, IL)
* Categorical data will be described as numbers and percentage
* Data will be explored for normality using Kolmogrov-smirnov test and Shapiro-wilk test
* Comparison between two groups for normally distributed numeric variables will be done by Mann-Whitney test. An equivalence limit will be tested.
* A P-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Data monitoring:

Monitoring The main supervisor is responsible of data monitoring if harms arise, interim analysis will be done.

Harms Any adverse effect like pain or even failure will be recorded, documented and treated.

Audit Auditing of the study design will be done by the evidence-based committee of the faculty of Oral and Dental medicine at Cairo University.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-55 years, are able to read and sign the informed consent document.
2. Patients who are physically and psychologically able to tolerate conventional restorative procedures.
3. Patients with no active periodontal or pulpal diseases and have teeth with good restorations.
4. Patients with complaints related to the esthetics in the upper or lower teeth (e.g. discoloration, fracture that does not involve more than 50% enamel loss, mild malposition)

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patient with fractured teeth of more than 50% enamel loss.
3. Patients with poor oral hygiene.
4. Patient with non-vital teeth.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
shade match | immediately after restoration delivery
  measured by Modified United States Public Health Service criteria (USPHS criteria). Score Alpha (A): matches tooth, Bravo (B): acceptable mismatch, Charlie (C): unacceptable mismatch

SECONDARY OUTCOMES:
marginal adaptation | immediately after restoration delivery
  measured by Modified United States Public Health Service criteria (USPHS criteria). Score Alpha (A): no catch with explorer , Bravo (B):explorer catches , Charlie (C): explorer penetrates
patient satisfaction | immediately after restoration delivery
  measure by Questionnaire (Scores are non-acceptable, acceptable, good and excellent).